CLINICAL TRIAL: NCT04298268
Title: Clinical Performance Investigation of the CUSA® Clarity Ultrasonic Surgical Aspirator System for Soft Tissue Removal During Urological and General Surgery
Brief Title: The CUSA Clarity Soft Tissue Removal Study
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-CUSATR-001
Record Dates: First submitted 2020-02-18; First posted 2020-03-06 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Benign, Malignant Tumors or Other Soft Tissue Removal; Nephrectomy or Partial Nephrectomy With Parenchyma Removal
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: CUSA Clarity Ultrasonic Surgical Aspirator System use — Assessment of the CUSA® Clarity Ultrasonic Surgical Aspirator System use during urological or general surgery for soft tissue removal

SUMMARY:
To investigate the clinical performance and surgeon preferences of the CUSA® Clarity Ultrasonic Surgical Aspirator System for soft tissue removal during surgical procedures. This will be evaluated through the effectiveness of soft tissue removal per surgeon assessment and Incidence of Adverse Device Effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject requires removal of soft tissue with an ultrasonic aspirator during urological or general surgery
* Subject is an appropriate candidate to receive use of the CUSA® Clarity Ultrasonic Surgical Aspirator System product for soft tissue removal during surgery, per the study surgeon
* Subject signed the IRB/EC-approved informed consent form demonstrating that the subject is willing and able to participate in this clinical study and to comply with all study procedures, if applicable.

Exclusion Criteria:

* Subject is currently pregnant or plans to become pregnant prior to the study index surgery
* Subject has any significant medical condition that in the opinion of the investigator will interfere with protocol evaluation and participation
* Subject's surgical plan includes utilizing CUSA® Clarity Ultrasonic Surgical Aspirator System for the removal of uterine fibroids
* Subject is a prisoner or member of a different vulnerable population that should not be included in the study per the investigator or ethics committee.
* Intra-operative exclusion criteria : Surgeon does not utilize the CUSA® Clarity Ultrasonic Surgical Aspirator System for soft tissue removal during surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient requiring removal of soft tissue with an ultrasonic aspirator during urological or general surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness of soft tissue removal per surgeon assessment. | During the surgery
  Multifactorial 5-point Likert scale (1 (worst) to 5 (best))

CONTACTS AND LOCATIONS:
Overall Officials: Jason Marzuola, Study Director — Integra LifeSciences
Locations (5):
- Klinikum Dortmund, Dortmund, Germany
- Italy (4):
  - Niguarda Hospital, Milan
  - ISMETT, Palermo
  - Hopital Gemelli U.O.C. Chirurgia Generale ed Epatobiliare, Roma
  - Policlinico Universitario Agostino Gemelli, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Accardo C, Gruttadauria S, Decarlis L, Agnes S, Schmeding M, Avolio AW, Buscemi V, Ardito F, Kienlein S, Mbuvi PM, Giuliante F. The CUSA Clarity Soft Tissue Removal Study: Clinical Performance Investigation of the CUSA Clarity Ultrasonic Surgical Aspirator System for Soft Tissue Removal During Liver Surgery. J Laparoendosc Adv Surg Tech A. 2024 Feb;34(2):99-105. doi: 10.1089/lap.2023.0467. Epub 2024 Jan 31. PMID 38294895